CLINICAL TRIAL: NCT06432023
Title: Multi-signal Analysis of the Composition and Movement of Fluid in Various Cerebral Compartments in Healthy Subjects and Subjects With White Matter Pathology
Brief Title: Imaging - Clinical Evaluation of Altered Nervous System Drainage
Acronym: I-CLEANED
Status: Recruiting | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1022
Record Dates: First submitted 2024-05-15; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Neuroinflammation; Autism Spectrum Disorder
Keywords: magnetic resonance imaging; autism spectrum disorder; white matter disease; glymphatic system; brain waste clearance
MeSH Terms: conditions — Neuroinflammatory Diseases; Autism Spectrum Disorder; Leukoencephalopathies | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: patients with white matter hyperintensities, patients with enlarged perivascular spaces, Focus will be on patients with a clinical diagnosis of muscular dystrophy or autism spectrum disorder or traumatic brain injury.
  Interventions: Diagnostic Test: Magnetic resonance imaging
- Controls: Patients who need a diagnostic scan but do not carry a diagnosis of psychomotor or cognitive impairment or without a history of TBI and tumors. No white matter hyperintensities.
  Interventions: Diagnostic Test: Magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging — Diagnostic and research scanning using magnetic resonance imaging.

SUMMARY:
The current study aims to evaluate the aspects of perfusion, fluid diffusivity in the interstitium and the T1 and T2 signal of the PVS and WMH. The current study has the following objectives: a) evaluate the perfusion aspects using the gadolinium-based contrast medium of brain tissues in the short term; b) the direction of flow of fluids at very low speed in the white matter using the DTI sequences configured for this purpose; c) T1-mapping of the lesions of interest.

The expected results will help us understand two aspects of neurofluid dynamics: a) how the fluid moves within the central nervous system in the first minutes after the injection of the tracer (in our case the gadolinium-based contrast medium) and b) what is the composition of the fluid within the PVS and WMH and how can investigators characterize them more accurately.

DETAILED DESCRIPTION:
Among the various indirect markers of altered drainage of neuroglial waste metabolites, there is the widening of the perivascular spaces (PVS) and the presence of white matter signal alterations.

An increase in the number of PVS and their enlargement could represent an indirect marker of obstruction to the drainage of fluids and solutes along the arterial wall at the level of the white matter. This obstruction would also be the basis of tissue hypoxia resulting in the formation of areas of signal hyperintensity in the white matter (White Matter Hyperintensities, WMH) often observed in patients with neurodegenerative diseases and small vessel disease.

It is currently unclear what the main drainage route of brain waste metabolites is. Surely there are at least two.

The glymphatic theory proposes the entry of the cerebrospinal fluid (CSF) from the subarachnoid space towards the brain parenchyma in a centripetal direction and exit of the metabolic waste along the perivenous spaces. The drainage of metabolic waste could also be explained by the more recent "intramural periarterial drainage" (IPAD) theory which shows elimination along the arterial walls in a centrifugal direction.

In magnetic resonance imaging (MRI), the study of solute drainage requires a dynamic evaluation, which is able to evaluate the temporal movement of a tracer. There are several MRI techniques, already described in the literature, which can be used to obtain information relating to perfusion processes and the coupling of neuronal and vascular activity in different brain areas.

The circulation of CSF is well known, which is produced largely at the level of the choroid plexuses and is then partly reabsorbed by the arachnoid granulations at the level of the subarachnoid space. Recent studies demonstrate that the CSF re-enters the brain parenchyma in a centripetal manner, crossing the thickness of the gray matter and then the white matter. This movement is regulated by various factors, and in particular by the activity of the smooth muscle cells of the arterial walls, the aquaporin 4 receptors (water channels) and by the chemical-physical properties of the extracellular matrix in the extracellular space.

ELIGIBILITY:
Inclusion Criteria:

* patients with white matter lesions and/or enlarged perivascular spaces

Exclusion Criteria:

* have contraindications to the use of contrast medium;
* are clinically unstable patients and prolonged sedation is inappropriate
* have tumors
* contraindications to perform MR.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with obvious white matter disease on T2 and FLAIR sequences will be included in this study. In particular patients with recent diagnosis of autism spectrum disorder, traumatic brain injury, Steinert's muscular dystrophy will be included.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Perivascular space count | once at recruitment
  Number and distribution of enlarged perivascular spaces
Volume of parasagittal dura | once at recruitment
  correlation of parasagittal dura and perivascular count
fMRI signal during sedation | once at recruitment
  effect of sedation on BOLD signal

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Institute IRCCS E. Medea, Bosisio Parini, Lecco, Italy

IPD SHARING:
Plan to Share IPD: Undecided